CLINICAL TRIAL: NCT03369015
Title: Effect of D-amphetamine on Reward Functioning
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Scott Lane, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HSC-MS-17-0604
Record Dates: First submitted 2017-11-20; First posted 2017-12-11 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Anhedonia
Keywords: Reward Learning; Decision Making
MeSH Terms: conditions — Anhedonia | interventions — Dextroamphetamine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Placebo, then 10 mg d-amphetamine, then 20mg d-amphetamine (Experimental)
  Interventions: Drug: 10 mg d-amphetamine; Drug: 20mg d-amphetamine; Drug: Placebo
- Placebo, then 20 mg d-amphetamine, then 10mg d-amphetamine (Experimental)
  Interventions: Drug: 10 mg d-amphetamine; Drug: 20mg d-amphetamine; Drug: Placebo
- 10 mg d-amphetamine, then placebo, then 20mg d-amphetamine (Experimental)
  Interventions: Drug: 10 mg d-amphetamine; Drug: 20mg d-amphetamine; Drug: Placebo
- 10 mg d-amphetamine, then 20mg d-amphetamine, then placebo (Experimental)
  Interventions: Drug: 10 mg d-amphetamine; Drug: 20mg d-amphetamine; Drug: Placebo
- 20 mg d-amphetamine, then 10mg d-amphetamine, then placebo (Experimental)
  Interventions: Drug: 10 mg d-amphetamine; Drug: 20mg d-amphetamine; Drug: Placebo
- 20 mg d-amphetamine, then placebo, then 10mg d-amphetamine (Experimental)
  Interventions: Drug: 10 mg d-amphetamine; Drug: 20mg d-amphetamine; Drug: Placebo

INTERVENTIONS:
Drug: 10 mg d-amphetamine — 10 mg d-amphetamine dose given (double-blind) and behavioral tasks (EEfRT, PRT, ELT, CGT) administered.
Drug: 20mg d-amphetamine — 20 mg d-amphetamine dose given (double-blind) and behavioral tasks (EEfRT, PRT, ELT, CGT) administered.
Drug: Placebo — Placebo dose given (double-blind) and behavioral tasks (EEfRT, PRT, ELT, CGT) administered.

SUMMARY:
The purpose of this study is to establish the dose-response curve for therapeutic doses of d-amphetamine on tasks of motivation and reward learning in the same participants and to use d-amphetamine as a dopaminergic probe to test newer theories about the role of dopamine in reward-related decision-making.

ELIGIBILITY:
Inclusion Criteria:

- Healthy individuals

Exclusion Criteria:

* Individuals with a body mass index (BMI) <19 or >26, as this alters dosing requirements
* Individuals with high blood pressure, abnormal Electrocardiography (EKG), any medical condition requiring regular medication (except birth control), any other regular use of a drug or supplement with potentially hazardous interactions with d-amphetamine (e.g. St. John's wort), or any other medical contraindication to amphetamine administration as determined by our study physician
* Individuals who report no prior experience with recreational drugs of any kind (including alcohol), or who report a previous adverse reaction to amphetamine
* Individuals with a current Diagnostic and Statistical Manual of Mental Disorders-V (DSM-V) Axis I diagnosis, excluding mild Substance Use Disorders (≤ 3 symptoms)
* Individuals with a lifetime history of moderate to severe Substance Use Disorder (≥ 4 symptoms), mania or psychosis.
* Women who are pregnant.
* individuals smoking more than 10 cigarettes per week will also be excluded, to avoid confounding the effects of nicotine withdrawal with the effects of the study drugs/procedures, as participants will not be allowed to smoke during the sessions.
* individuals with less than a high-school level of education or fluency in English will be excluded as our questionnaires require high-school level fluency in English, and have not been translated and validated in other languages.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Reward motivation as assessed by the Effort Expenditure for Reward Task (EEfRT) | about 100 minutes to 140 minutes after receiving drug at 1st, 2nd, and 3rd study session
  A measure of effort-based decision-making in humans, the Effort Expenditure for Reward Task (EEfRT), will be used. The EEfRT requires participants to choose between a low-effort, low reward task vs a high-effort, high reward task. Willingness to exert effort, or reward motivation, is measured by taking the average number of hard task choices from the first 50 trials.
Reward learning as assessed by the Probabilistic Reward Task (PRT) | about 100 minutes to 140 minutes after receiving drug at 1st, 2nd, and 3rd study session
  The Probabilistic Reward Task (PRT), which uses a signal detection paradigm, will be used to measure response bias towards rewarded stimuli.

SECONDARY OUTCOMES:
Reward learning as assessed by the Effort Learning Task (ELT) | about 100 minutes to 140 minutes after receiving drug at 1st, 2nd, and 3rd study sessions
  The novel Effort Learning Task (ELT) will be used, in which participants learn to associate abstract shapes with reward, loss, high effort and low effort outcomes, to examine the effect of dopaminergic stimulation on reward learning. Learning rates are determined for each symbol, and trial-wise learning curves are calculated as metrics of reward learning.
Level of influence of counterfactual information on later decision-making, as measured by the Counterfactual Gambling Task (CGT) | about 100 minutes to 140 minutes after receiving drug at 1st, 2nd, and 3rd study session
  Striatal dopamine is involved in signalling counterfactual information, i.e. encoding differences between the value of actual outcomes and hypothetical outcomes of alternative choices. The CGT is a gambling task used to assess the relationship between choice factors (available options, expected value, and outcomes) on self-reported measures of momentary happiness and regret. Participants complete a gambling task and are informed of their outcome and of the counterfactual outcome (i.e. hypothetical outcome had the participant selected another option). With this task, the degree to which participants make choices to avoid potential regret can be estimated.
Mood state as assessed by the Profile of Mood States (POMS) | 15 minutes before receiving drug and 30, 90, 180, and 210 minutes after receiving drug at 1st, 2nd, and 3rd study sessions
  The effect of d-amphetamine on mood state will be assessed throughout sessions and will be used as a manipulation check.
Subjective effects of drug as assessed by the Drug Effects Questionnaire (DEQ) | 15 minutes before receiving drug and 30, 90, 180, and 210 minutes after receiving drug at 1st, 2nd, and 3rd study sessions
  The pharmacodynamics of d-amphetamine will be assessed throughout the study and will be used as a manipulation check.

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Lane, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States